CLINICAL TRIAL: NCT06670196
Title: A Randomized, Open-Label, Multicenter, Phase III Clinical Study of SKB264 in Combination With Osimertinib Versus Osimertinib Alone as First-Line Treatment for Patients With Epidermal Growth Factor Receptor (EGFR) Mutations, Locally Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of SKB264 in Combination With Osimertinib Versus Osimertinib in Patients With Epidermal Growth Factor Receptor (EGFR) Mutations, Locally Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅲ-15
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: SKB264; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 1:1 ratio to one of two intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKB264+Osimertinib (Experimental): Participants will receive SKB264 on Day 1 and Day 15 of each 4-week cycle, Osimertinib once-daily for each 4-week cycle.
  Interventions: Drug: SKB264; Drug: Osimertinib
- Osimertinib (Active Comparator): Participants will receive Osimertinib once-daily for each 4-week cycle.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: SKB264 — 4mg/kg, intravenous (IV) infusion
  Arms: SKB264+Osimertinib
Drug: Osimertinib — 80mg, QD

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of SKB264 in combination with osimertinib as first-Line treatment for patients with epidermal growth factor receptor (EGFR) mutations, locally advanced or metastatic non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a randomized, open-Label, multicenter, Phase 3 study to evaluate the efficacy and safety of SKB264 in combination with osimertinib versus osimertinib alone as first-line treatment for patients with EGFR mutations, locally advanced or metastatic non-squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years to ≤75 years at the time of signing the informed consent form (ICF), regardless of gender.
2. Histologically or cytologically confirmed non-squamous NSCLC that is locally advanced (stage IIIB/IIIC) or metastatic (stage IV) non-squamous NSCLC not eligible to radical surgery and/or radical radiotherapy.
3. No prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC.
4. Histologically or cytologically confirmed EGFR-sensitive mutations.
5. Tumor tissue samples obtained at or after the diagnosis of locally advanced or metastatic tumor are eligible.
6. At least one target lesion assessed by the investigator based on RECIST v1.1.
7. ECOG performance status score of 0 or 1 within 7 days prior to randomization.
8. Life expectancy ≥ 12 weeks.
9. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Histologically or cytologically confirmed presence of small cell lung cancer, neuroendocrine carcinoma, and carcinosarcoma components or squamous cell carcinoma components of more than 10%.
2. Subjects who have received prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC.
3. Subjects who have received any of the following therapies (including the adjuvant/neoadjuvant therapy):

   1. Targeted TROP2 therapy;
   2. Any drug therapy that targets topoisomerase I, including antibody-drug conjugates (ADCs).
4. Subjects with known meningeal metastases, brainstem metastases, spinal cord metastases and/or compression, active or central nervous system (CNS) metastase.
5. Other malignancies within 3 years prior to randomization.
6. Clinically significant abnormalities found on resting electrocardiogram (ECG)
7. Presence of any of cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors.
8. History of interstitial lung disease (ILD), drug-induced ILD, history of non-infectious pneumonitis requiring steroid treatment, current ILD or non-infectious pneumonitis.
9. Clinically severe lung injuries caused by lung diseases.
10. Unresolved toxicities from previous anti-tumor therapy to ≤ Grade 1 (based on NCI CTCAE v5.0) or the level specified in the inclusion and exclusion criteria.
11. Subjects who have received systemic corticosteroids > 10 mg/day of prednisone or other immunosuppressive agents within 2 weeks prior to randomization.
12. Known active pulmonary tuberculosis.
13. Known history of allogeneic organ transplant and allogeneic hematopoietic stem cell transplant.
14. Presence of active hepatitis B or hepatitis C.
15. Positive result of human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.
16. Known allergy to osimertinib, SKB264 or any of their components (including but not limited to polysorbate-20), history of severe hypersensitivity to other biologics.
17. Vaccination with live vaccines within 30 days prior to randomization, or planned vaccination with live vaccines during the study.
18. Women who are pregnant or breastfeeding.
19. Presence of local or systemic diseases caused by non-malignancies, or diseases or symptoms secondary to tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by Blinded Independent Central Review (BICR) | Randomization up to approximately 36 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Randomization up to approximately 49 months
  OS is defined as the time from randomization until the date of death due to any cause.
Progression-Free Survival (PFS) assessed by Investigator | Randomization up to approximately 36 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) | Randomization up to approximately 36 months
  ORR is defined as the percentage of patients who achieve complete response(CR) or partial response (PR), as assessed by BICR/investigator per RECIST 1.1
Disease control rate (DCR) | Randomization up to approximately 36 months
  DCR is defined as the percentage of patients who achieve CR, PR or stable disease (SD), as assessed by BICR/ investigator per RECIST 1.1
Duration of Response (DoR) | Randomization up to approximately 36 months
  DoR is defined as the time from the date of first documented CR or PR until date of documented disease progression per RECIST 1.1, as assessed by BICR/investigator or death due to any cause, whichever occurs first.
Time to Response (TTR) | Randomization up to approximately 36 months
  TTR is defined as the time from the date of randomization until the first documentation of CR or PR as assessed by BICR/investigator per RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China